## **INFORMED CONSENT FORMS**

# Official Title of the Study:

Forgetting Alcohol: A Double-blind, Randomized Controlled Trial Investigating Memory Inhibition Training in Young Binge Drinkers

NCT ID: not yet assigned

Date: February 5, 2019





University of Minho School of Psychology Research Center in Psychology (CIPsi) Psychological Neuroscience Laboratory Campus de Gualtar 4710-057 Braga Tel: +351 253 601 398

Research Project reference: NORTE-01-0145-FEDER-028672

Principal Investigator (PI) and Research Team: Dr. Eduardo López Caned (PI); Dra. Adriana

Sampaio e Dr. Alberto Crego

## **INFORMED CONSENT FORM**

### **COPY FOR THE PARTICIPANT**

| $\Box$ 1) I confirm I have read and understood the informative document that was delivered to me, with all the information regarding the study in which I am participanting, and that I had the opportunity to raise questions and doubts about it. |
|---|
| $\square$ 2) I confirm the research team had provide me clear answers to all my questions and doubts. |
| □3) I understand that I am free to leave the study at every moment, without justification, and without any consequences. |
| □4) I understand and agree that my personal identification data and the data obtained trhough the course of the research study will be kept in separate archives, therefore guaranteeing its safety, and that the team members with access to the data will respect their confidentiality. |
| □5) I, therefore, consint that my data are stored and/or exported to external databases in order to be analyzed, understading that, in any circumstance, information regarding my identity will not be disclosed. |
| □6) I understand that the presente study does not have a diagnostic purpose and, consequentely, I will not receive na individual report with my data/results. |
| □7) I consint to participate in the abovemnetioned study. |
| Participant name: |
| Researcher name: |
| Name of the person responsible for collecting this consent (if different from the researcher): |
| Date: Participant Code: |





University of Minho School of Psychology Research Center in Psychology (CIPsi) Psychological Neuroscience Laboratory Campus de Gualtar 4710-057 Braga Tel: +351 253 601 398

**Research Project reference**: NORTE-01-0145-FEDER-028672

Principal Investigator (PI) and Research Team: Dr. Eduardo López Caned (PI); Dra. Adriana

Sampaio e Dr. Alberto Crego

Date: .....

## **INFORMED CONSENT FORM**

#### **COPY FOR THE RESEARCHER**

| □1) I confirm I have read and understood the informative document that was delivered to me, with all the information regarding the study in which I am participanting, and that I had the opportunity to raise questions and doubts about it. |
|---|
| $\Box$ 2) I confirm the research team had provide me clear answers to all my questions and doubts. |
| $\Box$ 3) I understand that I am free to leave the study at every moment, without justification, and without any consequences. |
| □4) I understand and agree that my personal identification data and the data obtained trhough the course of the research study will be kept in separate archives, therefore guaranteeing its safety, and that the team members with access to the data will respect their confidentiality. |
| □5) I, therefore, consint that my data are stored and/or exported to external databases in order to be analyzed, understading that, in any circumstance, information regarding my identity will not be disclosed. |
| $\Box$ 6) I understand that the presente study does not have a diagnostic purpose and, consequentely, I will not receive na individual report with my data/results. |
| □7) I consint to participate in the abovemnetioned study. |
| Participant name: |
| Researcher name: |
| Name of the person responsible for collecting this consent (if different from the researcher): |

Participant Code: .....